CLINICAL TRIAL: NCT03160534
Title: Effect of Preoperative Exercise in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Pilot Trial
Brief Title: Effect of Preoperative Exercise in Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0472
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Pilot Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Preoperative exercise intervention
  Interventions: Other: preoperative exercise
- Control (No Intervention): Only measurements

INTERVENTIONS:
Other: preoperative exercise — Each intervention session contains a stretching part and aerobic training
  Arms: Intervention

SUMMARY:
This study evaluates the effect of preoperative exercise in patients undergoing a total knee arthroplasty.

DETAILED DESCRIPTION:
The objectives of this study were to investigate the effects of a single (9 sessions) prescription community based preoperative physical therapy in patients awaiting a Total Knee Arthroplasty, taking prognostic factors into account.

The investigators will use different outcome measures to evaluate any possible effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a Total Knee Arthroplasty
* Signed informed consent after being informed

Exclusion Criteria:

* Acute pain
* Weakness due to neurological problems
* Known or suspected non-compliance
* High BMI > 28
* Patellar residual subluxation
* High patellar height

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Stair climbing test | 5 minutes
  The stair climbing test (SCT) measures the time used to ascend and descend a flight of twelve steps. Patients are asked to complete the test as quickly as they felt safe and comfortable.

SECONDARY OUTCOMES:
Knee - Range of Motion | 2 minutes
  The range of motion of the knee will be assessed.
Tegner Activity Scale and Lysholm Score | 10 minutes
  The Lysholm score and the Tegner activity scale are widely used for assessing knee function and activity level after knee ligament injuries
Patient Global Impression of Change | 2 minutes
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment.
Risk of Discharge to a Rehabilitation Facility | 20 minutes
  Costs and duration of postoperative rehabilitation will be measured with help of a personal calendar. All participants will report on this calendar any post-acute care services after surgery, Costs of skilled nursing facilities, home health agencies, and inpatient rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
no there is not

REFERENCES:
- [Derived] Granicher P, Stoggl T, Fucentese SF, Adelsberger R, Swanenburg J. Preoperative exercise in patients undergoing total knee arthroplasty: a pilot randomized controlled trial. Arch Physiother. 2020 Aug 5;10:13. doi: 10.1186/s40945-020-00085-9. eCollection 2020. PMID 32774889